CLINICAL TRIAL: NCT03882255
Title: A Randomized, Double-blind, Parallel-group, 2-period, Placebo-controlled, Phase 1 Study to Investigate the Effects on Heart Rate, Blood Pressure, and Pharmacokinetic Interactions of the Up-titration Regimen of Ponesimod in Healthy Adult Subjects Receiving Propranolol at Steady State
Brief Title: A Study of Ponesimod in Healthy Adult Participants Receiving Propranolol at Steady State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108589; 2018-003550-24 (EudraCT Number); AC-058-117 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Period 1: Ponesimod (2 mg) (Experimental): Participants will receive a single dose ponesimod 2 milligram (mg) oral tablet under fed conditions on Day 1. Participants not fulfilling discontinuation criteria can continue to Treatment Period 2 after a washout period of at least 7 days and a maximum of 14 days.
  Interventions: Drug: Ponesimod dose range (2 - 20 mg)
- Treatment Period 2:Ponesimod, Propranolol, Placebo Propranolol (Experimental): Participants who do not fulfill any of discontinuation criteria will be randomized to 1 of 2 Treatments (Treatment A or B) on Day 1. Treatment A: up-titration regimen of ponesimod (2mg-20mg) once daily from Day 5 to Day 19 plus placebo propranolol once daily from Day 1 to Day 19; Treatment B: up-titration regimen of ponesimod (2mg-20mg) once daily from Day 5 to Day 19 plus 80 mg propranolol once daily from Day 1 to Day 19.
  Interventions: Drug: Ponesimod dose range (2 - 20 mg); Drug: Placebo Propranolol; Drug: Propranolol 80 mg

INTERVENTIONS:
Drug: Ponesimod dose range (2 - 20 mg) — Participants will receive ponesimod oral tablet at a dose of 2 mg in Treatment period 1 and as an up-titrating regimen (dose range: 2mg-20mg) in Treatments period 2.
Drug: Placebo Propranolol — Participants will be administered placebo propranolol oral capsule from Day 1 to Day 19 in Treatment A of Treatment period 2.
  Arms: Treatment Period 2:Ponesimod, Propranolol, Placebo Propranolol
Drug: Propranolol 80 mg — Participants will receive propranolol 80 mg long acting oral capsule from Day 1 to Day 19 in Treatment B of Treatment period 2.
  Arms: Treatment Period 2:Ponesimod, Propranolol, Placebo Propranolol

SUMMARY:
The primary purpose of this study is to evaluate the effect of the up-titration regimen of ponesimod on heart rate (HR) and other electrocardiogram (ECG) parameters when administrated to healthy adult participants receiving propranolol at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure (SBP) 90 to 140 millimeters of mercury (mmHg) and diastolic blood pressure (DBP) 50 to 90 mmHg measured on the right arm in supine position after at least 5 minutes rest in the supine position at screening, on Day 1 of the Treatment Period 1, and on Day -2 of Treatment Period 2
* Body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2 ) (inclusive) at screening and body weight not less than 50.0 kg
* 12-lead safety electrocardiogram (ECG) without clinically relevant abnormalities at screening, on Day 1 of the Treatment Period 1, and on Day-2 of Treatment Period 2, including:

  1. QT interval corrected for heart rate using the Fridericia correction (QTcF) of less than or equal to (=<) 450 millisecond (ms) for male participants and =< 470 ms for female participants
  2. Heart rate (HR) 55 to 100 Beats per minute (bpm) (inclusive)
  3. QRS interval less than (<) 120 ms
  4. PR interval =< 200 ms
  5. ECG morphology consistent with healthy cardiac conduction and function
* Female participant must have a negative highly sensitive serum (beta human chorionic gonadotropin [beta- hCG]) pregnancy test at screening and a negative urine pregnancy test on Day 1 of Treatment Period 1 and Day 2 of Treatment Period 2
* Negative results from urine drug screen at screening, on Day -1 of Treatment Period 1, and on Day -2 of Treatment Period 2

Exclusion Criteria:

* Any cardiac condition or illness (including ECG abnormalities) with a potential to increase the cardiac risk of the participant based on medical history, physical examination, 12-lead safety ECG, or 24-hour Holter ECG at screening, including:

  1. 24-hour Holter ECG with clinically relevant abnormalities
  2. History or evidence of Atrioventricular (AV) block second degree or higher
  3. Any cardiac condition or illness (including ECG abnormalities based on standard 12-lead safety ECG or d- 24-hour Holter ECG) with a potential to increase the cardiac risk of the participant
* Family history of sick-sinus syndrome
* Hepatitis A antibody immunoglobulin M (IgM) positive, positive hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-hepatitis C virus [anti-HCV]) tests, or other clinically active liver disease at screening
* Known hypersensitivity to any excipients of the ponesimod drug formulation (lactose, microcrystalline cellulose, povidone, sodium lauryl sulfate, croscarmellose sodium, colloidal anhydrous silica, magnesium stearate, opadry II brown), or lactose
* History of significant propranolol side effects or known hypersensitivity to propranolol or to any of its excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Maximum Decrease from Baseline in Mean Hourly Heart Rate (HR) (Emax HR) on Day 5 | Baseline and Day 5
  Emax HR is defined as the maximum decrease from baseline in mean hourly HR.
Maximum Decrease from Baseline in Mean Hourly Heart Rate (HR) (Emax HR) on Day 19 | Baseline and Day 19
  Emax HR is defined as the maximum decrease from baseline in mean hourly HR.
Minimum of the Mean Hourly HR for each day (HR nadir) on Day 5 | Day 5
  HR nadir will be defined as the minimum of the mean hourly HR for each day and will be summarized by descriptive statistics.
Minimum of the Mean Hourly HR for each day (HR nadir) on Day 19 | Day 19
  HR nadir will be defined as the minimum of the mean hourly HR for each day and will be summarized by descriptive statistics.

SECONDARY OUTCOMES:
Maximum Decrease from Baseline in Mean Hourly Heart Rate (HR) (Emax HR) on Days 4,16, and 19 | Baseline, Days 4, 16, and 19
  Emax HR is defined as the maximum decrease from baseline in mean hourly HR.
Minimum of the Mean Arterial Blood Pressure | Days 4, 5, 16, and 19
  Minimum of the Mean arterial blood pressure (MAP) will be assessed. The MAP will be derived from the systolic blood pressure (SBP) and diastolic blood pressure (DBP) for each participant at the same time point as follows: MAP = 1/3 SBP + 2/3 DBP.
Change from Baseline in Average Heart Rate | Baseline, Days 4, 5, 16, and 19
  Change from baseline in average heart rate on Days 4, 5, 16 and 19 will be assessed in Treatment Period 2.
Change from Baseline in Average PR Interval | Baseline, Days 4, 5, 16, and 19
  Change from baseline in PR interval on Days 4, 5, 16 and 19 will be assessed in Treatment Period 2. PR intervals will be derived from 12-lead safety electrocardiogram (ECG).
Maximum Observed Plasma Analyte Concentration (Cmax) of Ponesimod | Days 5, 9 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose)
  Cmax is defined as maximum observed plasma analyte concentration.
Maximum Observed Plasma Analyte Concentration (Tmax) of Ponesimod | Days 5, 19 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose)
  Tmax is defined as maximum observed plasma analyte concentration.
Area Under the Plasma Analyte Concentration-Time Curve (AUC [0-24]) of Ponesimod | Day 5 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 Hours postdose)
  (AUC [0-24]) is defined as area under the plasma analyte concentration-time curve (AUC) from time 0 to 24 hours postdose, calculated by linear-linear trapezoidal summation.
Trough Plasma Analyte Concentration (Ctrough) of Ponesimod | Day 19 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose)
  (Ctrough) is defined as observed analyte concentration just prior to the beginning of a dosing interval.
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Day 19 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose)
  The AUCtau is the measure of the plasma analyte concentration from time zero to end of dosing interval. AUC during a dosing interval (τ) at steady state, calculated by linear-linear trapezoidal summation.
Maximum Observed Plasma Analyte Concentration (Cmax) of Propranolol and 4 hydroxypropranolol | Days 4, 5, and 19 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose)
  Cmax is defined as maximum observed plasma analyte concentration.
Maximum Observed Plasma Analyte Concentration (Tmax) of Propranolol and 4 hydroxypropranolol | Days 4, 5, and 19 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose)
  Tmax is defined as maximum observed plasma analyte concentration.
Trough Plasma Analyte Concentration (Ctrough) of Propranolol and 4 hydroxypropranolol | Days 4, 5, and 19 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose)
  (Ctrough) is defined as observed analyte concentration just prior to the beginning of a dosing interval.
Area Under the Curve from Time Zero to End of Dosing Interval (AUCtau) of Propranolol and 4 hydroxypropranolol | Days 4, 5, and 19 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose)
  The AUCtau is the measure of the plasma analyte concentration from time zero to end of dosing interval. AUC during a dosing interval (τ) at steady state, calculated by linear-linear trapezoidal summation.
Total apparent Oral Clearance of Propranolol | Days 4, 5, and 19 (Predose; 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours postdose)
  Total apparent clearance is defined as total apparent oral clearance at steady state, calculated as dose/AUC (tau).
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Approximately 2.5 months
  An adverse event is any adverse change, that is, any unfavorable and unintended sign, including an abnormal laboratory finding, symptom, or disease, that occurs in a participant during the course of the study, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (1):
- SGS Clinical Pharmacology Unit (located in ZNA Stuivenberg), Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency